CLINICAL TRIAL: NCT01785043
Title: Differences in Endothelial Function Amongst Sitagliptin and Liraglutide Users: A Randomized, Open-label, Parallel-group and Active Controlled Trial
Brief Title: Differences in Endothelial Function Amongst Sitagliptin and Liraglutide Users
Acronym: LAED001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anna Cruceta (Other)
Responsible Party: Sponsor-Investigator, Anna Cruceta, Project manager Clinical Trials Unit, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAED001
Record Dates: First submitted 2013-01-07; First posted 2013-02-06 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: DIABETES Mellitus Type 2 Not Well Controlled
Keywords: DIABETES Mellitus Type 2; Difficult control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental): Liraglutide will be administered once a day by subcutaneous injection (under the skin) in the abdomen, thigh, or upper arm. It will be given independently of meals and preferably at the same each day. The starting dose will be 0.6 mg. After one week, the dose will be increased to 1.2 mg, and then it will be increased to 1.8 mg one week later to achieve better control of blood glucose. When Liraglutide is added to existing treatment containing metformin, as it is our scenario, the dose of metformin does not have to be changed.
  Interventions: Drug: Liraglutide
- Sitagliptin (Active Comparator): Sitagliptin will be administered once daily at a 100 mg dose. When Sitagliptin is used in combination with metformin, as it is our scenario, the dose of metformin should be maintained. If a dose of Sitagliptin is missed, it should be taken as soon as the patient remembers. A double dose should not be taken on the same day.
  Sitagliptin will be used daily during the study period of 12 weeks.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Liraglutide — Liraglutide is available if pre-filled pens (6 mg/ml) as a solution for injection (Victoza®). One ml of solution contains 6 mg of Liraglutide (human glucagon-like peptide-1 analogue produced by recombinant DNA technology in Saccharomyces cerevisiae). One pre-filled pen contains 18 mg Liraglutide in 3 ml.
  Other Names: Victoza®
  Arms: Liraglutide
Drug: Sitagliptin — Sitagliptin is available in 100 mg film-coated tablets (Januvia®). Each tablet contains sitagliptin phosphate monohydrate, equivalent to 100 mg sitagliptin.
  Other Names: Januvia
  Arms: Sitagliptin

SUMMARY:
Differences in endothelial function amongst Sitagliptin and Liraglutide Users. A randomized, open-label, parallel-group and active controlled trial

DETAILED DESCRIPTION:
Randomized, open-label, parallel-group, active controlled, phase IV study to assess the efficacy and safety of a 3 month treatment period with Liraglutide to Sitagliptin in type 2 diabetes patients not well controlled at the maximum tolerated dose of metformin.The study has been designed with a random design as it is one of the most important techniques for avoiding bias in clinical trials. The study will follow a parallel group, open-label design as liraglutide is administered by subcutaneous injection and sitagliptin orally in tablets. A double-dummy design has been rejected because it is highly complicated in a phase IV study, and any bias of an open-label design has a lower impact on objective variables (as it is our primary endpoint) and it could be compensated with the proposed random design.Sitagliptin has been selected as the active control as it is one of the prescribed treatments for type 2 diabetes patients not well controlled at the maximum tolerated dose of metformin.

The study objectives will be assessed after 3 months of therapy as it is considered a suitable timing for identifying short-term changes on flow-mediated vasodilation

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)
2. Male or female patients between 45 and 65 years old
3. Pre-existing type 2 diabetes with HbA1c between 7.0 and 9.5%
4. Triglycerides >1.68 mmol/L
5. HDL cholesterol <1.29 mmol/L in women and <1.04 mmol/L in men
6. Systolic blood pressure (SBP) <130 mmHg and diastolic blood pressure (DBP) <85 mmHg or treatment with antihypertensive agents

Exclusion Criteria:

1. Known or suspected hypersensitivity to trial product(s) or related products
2. Previous participation in this trial. Participation is defined as being randomised.
3. Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive, or males who are sexually active and not surgically sterilised, who or whose partner are not using adequate contraception
4. Moderate or severe renal dysfunction (creatinine clearance <60 ml/min)
5. Previous type 2 diabetes treatment apart from metformin or insulin
6. Current smoker or history of smoking within 6 months prior to screening.
7. Evidence of overt cardiovascular disease, (documented coronary heart disease, class II-IV congestive heart failure, cerebrovascular disease, or peripheral vascular disease).
8. Caffeine intake within 24 hours of endothelial function measurements.
9. Use of any drug with known clinically significant sympathetic or parasympathetic effects, as determined by the Investigator.
10. Initiation or change (dose or treatment regimen) in concomitant blood pressure-lowering medication within 4 weeks prior to screening and throughout the day.
11. The receipt of any investigational medicinal product within 6 months prior to screening.
12. Presence of cancer or other significant medical condition
13. Inability to follow verbal or written instructions

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Assess the effects on endothelial function of a three month treatment with Liraglutide compared to Sitagliptin. | 3months
  The primary objective is to assess the effects on endothelial function of a three month treatment with Liraglutide compared to Sitagliptin, assessed as the baseline corrected change in endothelial function by flow-mediated vasodilation (FMD) of the brachial artery at 3 months.

SECONDARY OUTCOMES:
The evaluation of other emerging potential cardiovascular risk factors | 3months
  1. Secondary objectives will include the evaluation of other emerging potential cardiovascular risk factors, such as oxidative stress markers, cytokines, and soluble cell adhesion molecules.
  2. The safety profile of both treatment groups will be also evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Ceriello, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain